CLINICAL TRIAL: NCT02950402
Title: Impact of California Dried Plums on Markers of Bone, Cardiovascular and Digestive Health
Brief Title: Dried Plums and Chronic Disease Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 843989
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Healthy, Postmenopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two Dried Plums per day (Experimental): Two Dried Plums per day is approximately 14 g.
  Interventions: Other: Two Dried Plums per day; Other: Six Dried Plums per day
- Six Dried Plums per day (Experimental): Six Dried Plums per day is approximately 42 g.
  Interventions: Other: Two Dried Plums per day; Other: Six Dried Plums per day

INTERVENTIONS:
Other: Two Dried Plums per day — Subjects will consume Two Dried Plums per day
Other: Six Dried Plums per day — Subjects will consume Six Dried Plums per day

SUMMARY:
This study evaluates whether the consumption of California dried plums can be beneficial to your health. Previous studies using dried plums have shown beneficial effects on bone and cardiovascular health. In addition the investigators hope to learn how dried plums might change your bowel habits, and if the carbohydrates in the plums are fermented in your digestive tract.

DETAILED DESCRIPTION:
The aging of the U.S. population presents a number of challenges, many of which that can be addressed through nutritional approaches. Postmenopausal women are particularly at-risk for a number of diseases such as osteoporosis (By 2020 it is estimated that 50 percent of women at 50 years and older will either suffer from or be at-risk of bone loss), and cardiovascular disease, the number one killer of postmenopausal women. Polyphenolic compounds in fruits and nuts have been the focus of extensive research regarding their potential to reduce risk for a number of chronic diseases. All fruits are not created equally, so determining if dried plums (Prunus domestica L.) have certain phytochemicals in amounts that promote health when consumed in realistic amounts is important. This demonstration is likely to impact market demand for dried plums. Indeed, favorable research on other California specialty crops (walnuts, almonds, strawberries, grapes) is a key strategy to help growers increase sales.

While hundreds of plum cultivars exist, with varying amounts of phenolic compounds, the process of drying results in high amounts on hydroxycinnamic acids, a family of compounds that have been shown, in animal models, to be protective of bone health by both reducing bone loss and improving bone growth. Hydroxycinnamic acids have also been proposed to improve vascular function by protecting the smooth endothelial lining of the blood vessels in animal models. Whether these encouraging observations also occur in humans is unknown. Therefore, the overall objective of this project is to conduct the first human study exploring the effects of California dried plums on markers of bone health and vascular function. Favorable results from this project will increase awareness of the unique benefits of dried plums for bone health and vascular health, two topics of great interest to aging baby boomers and other health-conscious consumers, both in the U.S. and internationally.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years of age
* Lack of menses in the last year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing participate in all study procedures
* BMI 18.5 - 34.9 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI < 18.5 kg/m2
* BMI ≥ 35 kg/m2
* Dislike or allergy for dried plums
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Self-reported use of oral cortisone or other immunosuppressive agents,
* Self-reported underlying neoplasia or immunological disease
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet • Alcohol consumption > 3 drinks/week (i.e. 1 bottle of beer, ½ glass of wine, and 1 shot of hard liquor)
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day for females
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and Stroke
* Self-reported Cushing's syndrome
* Self-reported chronic/routine high intensity exercise
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Use of multi-vitamin and mineral other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].

(using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);

* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

The following special populations will be excluded:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
C-telopeptide, beta-cross-linked (CTX), a marker of bone resorption | Change measures ("baseline and 2 weeks")
  To determine whether short-term (two weeks) intake of California dried plums will improve markers of bone health, as measured by a serum marker of bone remodeling called C-telopeptide, beta-cross-linked (CTX)

SECONDARY OUTCOMES:
Peripheral artery tonometry (PAT), a vascular function measure | Change measures ("baseline and 2 weeks")
  To determine whether short-term (two weeks) intake of California dried plums will improve vascular function, as measured using peripheral artery tonometry (PAT).
Breath hydrogen | Change measures ("baseline and 2 weeks")
  To determine the extent in which dried plum intake changes colonic fermentation products in dried plums.
Complete metabolic panel | Change measures ("baseline and 2 weeks")
  Blood analyses will include measurements of complete blood cell count, comprehensive metabolic panel, and lipid profile.
Body weight | Change measures ("baseline and 2 weeks")
  Body weight will be recorded at baseline and after two weeks of dried plum intake.
Blood pressure | Change measures ("baseline and 2 weeks")
  The baseline office blood pressure measurement will be obtained (3 measurements 5 minutes apart after a 15 minute rest).

IPD SHARING:
Plan to Share IPD: No